CLINICAL TRIAL: NCT00764673
Title: The 3DKnee™ System: A Post-Market Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Jane M. Jacob Ph.D., DJO Surgical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS - 703
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Results first posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-02

CONDITIONS: Osteoarthritis; Rheumatoid Arthritis; Post Traumatic Arthritis; Varus Deformity; Avascular Necrosis
MeSH Terms: conditions — Osteoarthritis; Arthritis, Rheumatoid; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Primary (Other): Post market study
  Interventions: Device: 3DKnee

INTERVENTIONS:
Device: 3DKnee — Subjects with knee osteoarthritis and willing to participate in the study

SUMMARY:
The purpose of this study is to evaluate the survivorship and efficacy of the Encore 3DKnee™ system in a group of patients who will receive the 3DKnee™ as a primary (first) orthopedic implant in the knee. Each knee will be designated as a separate subject and followed for a period of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* This must be a primary knee replacement on this knee.
* Have knee joint disease related to one or more of the following

  * degenerative joint disease, including osteoarthritis or traumatic arthritis
  * Avascular necrosis of the femoral condyles
  * Post-traumatic loss of joint configuration, particularly when there is patellofemoral erosion, dysfunction or prior patellectomy
  * Moderate valgus, varus, or flexion deformities
  * Rheumatoid arthritis
* Patient is likely to be available for evaluation for the duration of the study
* Able and willing to sign the informed consent and follow study procedures
* Patient is not pregnant
* Patient must be over 18 years of age

Exclusion Criteria:

* If there has been a total knee replacement on this knee in the past (no revisions allowed in study)
* Infection, or history of infection, acute or chronic, local or systemic
* Alcoholism or other addictions
* Muscular, neurological or vascular deficiencies which compromise the affected extremity
* Obesity
* Insufficient bone quality
* Loss of ligamentous structures
* High levels of physical activity
* Materials sensitivity
* Prisoner
* Mental conditions that may interfere with the patient's ability to give an informed consent or willingness to fulfill the study requirements
* Patient is pregnant
* Is younger than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2006-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McAllister, M.D., Principal Investigator — St. Peter's Bone and Joint Surgery
Locations (1):
- St. Peter's Bone & Joint Surgery, City of Saint Peters, Missouri, United States

REFERENCES:
- See also: Sponsor Company home page — http://www.djosurgical.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary 3DKnee Implant: Subjects who require a knee implant that have not previously had a knee replacement in the operative knee.
Period: Overall Study
Arm/Group | Primary 3DKnee Implant
Started | 71
Completed | 59
Not Completed | 12
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 6
Not completed — Revision of Device | 2

BASELINE CHARACTERISTICS:
Arm/Group | Primary 3DKnee Implant
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 69 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 71
Operated Knee [Number; unit: participants] — Affected knee which received the implant
  participants
    Right knee | 36
    Left knee | 35
Primary Diagnosis [Number; unit: participants] — Physician diagnosis of indication for receiving a total knee implant.
  participants
    Osteoarthritis | 69
    Varus deformity | 1
    Post-traumatic arthritis | 1

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score Evaluation
Description: The Knee Society Score includes a knee rating and function score. This evaluation covers the knee rating score with three main parameters of pain, stability and range of motion and that flexion contracture, extension lag and misalignment should be dealt with as deductions. Thus, 100 points will be obtained by a well-aligned knee with no pain, 125 degrees of motion, and negligible anteroposterior and mediolateral instability. 50 points are allotted for pain, 25 for stability, and 25 for range of motion. Grading for KS Score: Excellent (90-100), Good (80-90), Fair (70-79) and Poor (<70).
Time Frame: 2 year
Population: The number of subjects who completed their 2 year visit.
Measure: Mean (Standard Deviation); unit: Average Knee Rating Score
Arm/Group | Primary 3DKnee Implant
Number analyzed (Participants) | 59
Average Knee Rating Score | 82.9 (25.7)

2. Primary Outcome: Knee Society Function Score
Description: The Knee Society Score includes a knee rating and function score. Patient function considers only walking distance and stair climbing, with deductions for walking aids. The maximum function score, which is also 100, is obtained by a patient who can walk an unlimited distance and go up and down stairs normally. Walking ability is expressed in blocks (approximately 100 meters). Stair climbing is considered normal if the patient can ascend and descend stairs without holding a railing. A score of > or = to 60 on the function score is considered success.
Time Frame: 2-year
Population: The number of subjects who completed their 2 year visit and had available data to collect for this evaluation.
Measure: Mean (Standard Deviation); unit: Average Knee Function Score
Arm/Group | Primary 3DKnee Implant
Number analyzed (Participants) | 54
Average Knee Function Score | 76.6 (20.0)

3. Secondary Outcome: Oxford Knee Score
Description: Questionnaire on the perceptions of patients about a total knee replacement. Score between 0 and 48 where: 0 to 19 may indicate severe knee arthritis, 20 to 29 may indicate moderate to severe knee arthritis, 30 to 39 may indicate mild to moderate knee arthritis and 40 to 48 may indicate satisfactory joint function.
Time Frame: 2-year
Population: The number of subjects who completed an Oxford Knee score questionnaire at the 2 year visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Primary 3DKnee Implant
Number analyzed (Participants) | 59
Units on a scale | 36.3 (14.1)

4. Primary Outcome: Number of Participants With >2mm Wide at the Bone/Cement Interface or a >3 Degree or >3 mm Migration (Shift) of the Component.
Description: Radiographic failure is defined as a complete radiolucent line > 2mm wide at the bone/cement interface or a >3 degree or >3 mm migration (shift) of the component.
Time Frame: 2-year
Population: The number of subjects who came in for a 2 year visit and completed the x-ray portion of the evaluation.
Measure: Number; unit: participants
Arm/Group | Primary 3DKnee Implant
Number analyzed (Participants) | 59
participants | 0

5. Primary Outcome: Safety Assessment
Description: Number of device related adverse events and device failures at the 2 year time frame.
Time Frame: 2-year
Population: All subjects in the study were evaluated for adverse events.
Measure: Number; unit: Events
Arm/Group | Primary 3DKnee Implant
Number analyzed (Participants) | 71
Events
  Revisions of device | 2
  Number of device related adverse events | 18
  Total number of operative site events | 40

ADVERSE EVENTS:
Arm/Group | Primary 3DKnee Implant
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 62/71
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primary 3DKnee Implant (N=71)
Anemia (Blood and lymphatic system disorders) | 5 (5)
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 8 (8)
Brain disorder (Nervous system disorders) | 5 (5)
Device Instability (Surgical and medical procedures) | 3 (3) — 3DKnee device became loose.
Diabetes (Endocrine disorders) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Edema (Blood and lymphatic system disorders) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (5)
Heart Complications (Cardiac disorders) | 5 (5)
Wound infection, rash and/or redness (Infections and infestations) | 13 (13)
Kidney disorder (Renal and urinary disorders) | 2 (2)
Nausea (Injury, poisoning and procedural complications) | 2 (2)
Numbness (Nervous system disorders) | 6 (7)
Pain (Musculoskeletal and connective tissue disorders) | 38 (58)
Swelling (Vascular disorders) | 11 (12)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Urinary Tract Infection (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less